CLINICAL TRIAL: NCT05556317
Title: Effect of Resistive Exercise on Plasma Estradiol , Sleep Quality and Insomnia in Post Menopausal Women
Brief Title: Effect of Resistive Exercise on Insomnia in Post Menopausal Women
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Esraa Fikry Massoud Yamani, esraa fikry massoud yamani, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/003873
Record Dates: First submitted 2022-09-23; First posted 2022-09-27 (Actual); Last update posted 2022-09-27 (Actual); Status verified 2022-09

CONDITIONS: Sleep Disturbances and Insomnia
Keywords: Resistive exercise, insomnia, post menopausal women
MeSH Terms: conditions — Parasomnias; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: Resistive exercise on insomnia
Who Masked: Participant, Outcomes Assessor
Masking Description: Random generator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Receive advices to reduce insomnia
  Interventions: Behavioral: Resistive exercise
- Group B (Active Comparator): Receive advices and resistive exercise
  Interventions: Behavioral: Resistive exercise

INTERVENTIONS:
Behavioral: Resistive exercise — advices and resistive exercise

SUMMARY:
the aim of this study is to investigate the efficacy of resistive exercise on insomnia in post menopausal women

DETAILED DESCRIPTION:
Insomnia is a prevalent condition in post menopausal women.resistive exercise might play an important role in insomnia.this trial has two groups ;one will receive advices and the second will receive advices and resistive exercise for four week

ELIGIBILITY:
Inclusion Criteria:

1. age from 50 to 65 years
2. non smokers
3. BMI 25:29.9
4. post menopausal women suffer from insomnia

Exclusion Criteria:

1. post menopausal women suffer from any medical problems lead to sleep disturbance and insomnia
2. women on hormone replacement therapy
3. those with diagnosed osteoporosis

Ages: 50 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Post menopausal women
Enrollment: 56 (Estimated)
Dates: Start 2022-09-30 (Estimated); Primary Completion 2022-11-01 (Estimated); Study Completion 2022-11-15 (Estimated)

PRIMARY OUTCOMES:
Pittsburgh sleep quality index | Four week
  To determine sleep quality

SECONDARY OUTCOMES:
Insomnia severity index | Four week
  To determine insomnia

OTHER OUTCOMES:
Plasma estradiol | Four week
  To determine level of plasma estradiol

CONTACTS AND LOCATIONS:
Locations (1):
- Professor of physical therapy, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes